CLINICAL TRIAL: NCT06270979
Title: Feasibility and Usability of Intrinsic Capacity Monitoring With an Integrated Data Eco-System for Healthy Ageing, and Its Association With Health Outcomes in Older Patients Undergoing Rehabilitation and in Older Nursing Home Residents.
Brief Title: Intrinsic Capacity and Functional Ability Monitoring With an Integrated Data Eco-System for Healthy Ageing.
Acronym: ISHA
Status: Not yet recruiting | Type: Observational
Sponsor: Prof. Ivan Bautmans (Other)
Collaborators: Leiehome vzw (Unknown); University Hospital, Antwerp (Other); Universiteit Antwerpen (Other); INNOVIRIS (Unknown); AAL (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Ivan Bautmans, Professor, Vrije Universiteit Brussel
Organization: Vrije Universiteit Brussel (Other)
Other Study IDs: ISHA
Record Dates: First submitted 2024-01-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Frailty
Keywords: Self-monitoring; Intrinsic capacity; Prevention
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Leiehome vzw: Participant recruitment entails including persons aged 65 years or older living in an assisted housing or a nursing home.
  Interventions: Device: ISHA
- University Hospital Antwerp/University of Antwerp: Participant recruitment entails including persons aged 65 years or older undergoing rehabilitation at University Hospital Antwerp.
  Interventions: Device: ISHA

INTERVENTIONS:
Device: ISHA — Participants will be provided with an Eforto® device and ISHA mobile application to self-monitor intrinsic capacity for 4 months (if needed with assistance by an (in)formal caregiver).

SUMMARY:
In this study, 120 older adults (aged 65 years or older) either patients undergoing rehabilitation or older nursing home residents will be provided with an Eforto® device and the eco-System for Healthy Ageing (ISHA) mobile application to self-monitor intrinsic capacity for 4 months (if needed with assistance by an (in)formal caregiver). Preferably, the participants will use their own smartphone because mitigating smartphone-use-related issues.

The aims of the study are:

1. to evaluate the usability and feasibility of self-monitoring intrinsic capacity by using the ISHA system in rehabilitation and nursing home settings.
2. to investigate if changes and variability in intrinsic capacity as measured with ISHA are related to changes in functional ability and quality of life.
3. to explore individual trajectories of intrinsic capacity with the ISHA system.

DETAILED DESCRIPTION:
Investigational device:

The ISHA digital eco-system (class IIa investigational medical device).

ISHA consists of 3 components:

1. An Eforto® device: a handheld grip work (GW) hardware device, composed of a rubber bulb, to be compressed by the user and plastic enclosure that holds the electronic components such as a pressure sensor, battery, and connectivity. A mouthpiece can be attached for respiratory capacity monitoring.

   The Eforto® system was developed based on approximatively 20 years of scientific research on handgrip muscle fatigability performed by the Frailty in Ageing research department (see https://fria.research.vub.be/) and in collaboration with top-level international partners.

   The Eforto® system allows self-assessment of muscle fatigability and self-perceived fatigue in older adults and functions as a monitoring tool for intrinsic capacity. It is a small device, easy to use, and suitable for home measurements as well as hospital settings. When used correctly, the measurements cause no discomfort and can be performed repeatedly. The Eforto® device connects to a smartphone application that provides verbal test instructions to the participant. The app will guide the participant during the test and automatically provide motivational cues via audio. The test results are aggregated and stored in a cloud platform where the researcher can manage subjects, access the test data and export it for further analysis.
2. Mobile application that ensures connectivity and collection of data from the Eforto® device and by which multiple guided tests for the locomotor (maximal grip strength, respiratory muscle strength, muscle fatigue resistance test & self-perceived fatigue questionnaire), sensory (hearing test (signal to noise technology) & vision test (rotating E test), cognitive (orientation test, object naming from description, animal naming & 10-words immediate and delayed recall), and psychological (resilience questionnaire) domains of intrinsic capacity can be completed. The app allows offline data collection and to synchronize with the third component, the remote monitoring platform. It serves as an interactive guidance and can be used by the subject/patient at home or assisted by a (formal or informal) caregiver.
3. The remote monitoring platform serves mainly as a dashboard for monitoring the older end-users. Its main purpose is to centralize and monitor the collected data.

Procedures:

The study will be approved by the institutional review board's and all participants will sign informed consent.

After informed consent is given, the eligibility assessment and T0 (baseline) measurements will take place. These measurements will be re-assessed after 2 months and 4 months.

During this test moments the participant will be asked to perform the ISHA-tests (intrinsic domains: vitality, locomotor, sensory, cognitive and psychological). Other tests that will be assessed are: anthropometry (body weight & height and waist & hip circumference), health status (medical history, Center for Epidemiologic Studies Depression scale (CES-D), Mini Mental State Examination (MMSE), fall incidents, hospital admissions, Mini Nutritional Assessment (MNA) and orthostatic test), Frailty (Fried Criteria), functional dependency tests (Montreal Cognitive Assessment (MOCA), basic activity of daily living (ADL) (Katz), instrumental ADL (Lawton) and Short Physical Performance Test (SPPB)), questionnaires (Sarcopenia Quality of life questionnaire (SarQol), Eq-5D-5L, International Physical Activity Questionnaire (IPAQ), health-economic questionnaire and general health questions) and technical problem/ usability, feasibility and expectations questionnaires. In the context of eligible check, the smartphone experiences and personal data e.g. sex, birth day date, living situation will be asked.

After an individual information session with training on the ISHA test battery and instructions for ISHA use in self-test mode, the participant will be instructed to perform the ISHA measurements for 4 months at their home (if needed with assistance by an (in)formal caregiver). Preferentially, the healthcare professional (occupational therapist, physical therapist, study nurse) will install the ISHA application on the smartphone of the participant. If during the individual information session, the participant is unable to correctly operate the ISHA tool, the healthcare professional will explore together with the participant whether a (informal or formal) caregiver could aid, and eventually the participant will be re-invited together with his/her informal caregiver for another information/training session. If correct use of the ISHA system by the participant and/or assistance by a caregiver is impossible, the participant will be excluded for further participation in the study.

The self-test measurements will be continued for 4 months or until withdrawal of the participant. The self-tests will be performed:

* weekly on 2 consecutive days per week for vitality capacity;
* once every two weeks for locomotor capacity, and
* once every month for sensory, cognitive, and psychological capacity.

The application will give a reminder to the participant every time he/she needs to do the ISHA measurements.

During the study, participants will be contacted every month by a researcher to register any changes in health situation as well as technical issues encountered during the self-testing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older.
* Patients living independently at home and undergoing rehabilitation, or older persons living in the residential care community (in a nursing home or in assisted housing).
* Being able to operate the basic functions of a smartphone (if needed with assistance by an informal caregiver): using a smartphone at least for calls, and minimum 1 other application.
* Understanding Dutch.

Exclusion Criteria: Being unable to participate in the assessments due to:

* Being unable to perform the physical (self)tests (e.g., unable to stand up or walk);
* Being unable to understand the test instructions;
* Functional disability of the dominant upper extremity (paresis/paralysis, tremor or recent surgery);
* Patients undergoing neurological rehabilitation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients undergoing rehabilitation and nursing home residents, all aged 65 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Potential technical problems of the ISHA system | Week 1
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 2
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 3
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 4
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 5
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 6
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 7
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 8
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 9
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 10
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 11
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 12
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 13
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 14
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 15
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Potential technical problems of the ISHA system | Week 16
  A checklist of potential technical problems (12 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Experiences with ISHA (usability, feasibility and acceptability outcome) | End of the study (week 16)
  An self-reported questionnaire (19 questions) based on the System Usability Scale (SUS). Options for answer: 1-5. 1 is 'Strongly disagree', 5 is 'Strongly agree'.

SECONDARY OUTCOMES:
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (gait speed; m/s) measured with SPPB | Baseline
  Mobility is assessed by the SPPB, including gait speed(m/s) via the 4-meter test(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (gait speed; m/s) measured with SPPB | 2 months
  Mobility is assessed by the SPPB, including gait speed(m/s) via the 4-meter test(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (gait speed; m/s) measured with SPPB | 4 months
  Mobility is assessed by the SPPB, including gait speed(m/s) via the 4-meter test(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (gait speed; m/s) measured with SPPB | Baseline
  Mobility is assessed by the SPPB, including gait speed(m/s) via the 4-meter test(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (gait speed; m/s) measured with SPPB | 2 months
  Mobility is assessed by the SPPB, including gait speed(m/s) via the 4-meter test(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (gait speed; m/s) measured with SPPB | 4 months
  Mobility is assessed by the SPPB, including gait speed(m/s) via the 4-meter test(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (balance) measured with SPPB | Baseline
  Mobility is assessed by the SPPB, including balance, measured via the balance test.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (balance) measured with SPPB | 2 months
  Mobility is assessed by the SPPB, including balance, measured via the balance test.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (balance) measured with SPPB | 4 months
  Mobility is assessed by the SPPB, including balance, measured via the balance test.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (balance) measured with SPPB | Baseline
  Mobility is assessed by the SPPB, including balance, measured via the balance test.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (balance) measured with SPPB | 2 months
  Mobility is assessed by the SPPB, including balance, measured via the balance test.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (balance) measured with SPPB | 4 months
  Mobility is assessed by the SPPB, including balance, measured via the balance test.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (5-times sit-to stand (s)) measured with SPPB | Baseline
  Mobility is assessed by the SPPB, including 5-times sit-to stand tests(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (5-times sit-to stand (s)) measured with SPPB | 2 months
  Mobility is assessed by the SPPB, including 5-times sit-to stand tests(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability (5-times sit-to stand (s)) measured with SPPB | 4 months
  Mobility is assessed by the SPPB, including 5-times sit-to stand tests(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (5-times sit-to stand (s)) measured with SPPB | Baseline
  Mobility is assessed by the SPPB, including 5-times sit-to stand tests(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (5-times sit-to stand (s)) measured with SPPB | 2 months
  Mobility is assessed by the SPPB, including 5-times sit-to stand tests(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability (5-times sit-to stand (s)) measured with SPPB | 4 months
  Mobility is assessed by the SPPB, including 5-times sit-to stand tests(s).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with MoCa (0-30/30, the higher the better cognition) | Baseline
  Cognition will be assessed by the MoCa(0-30/30), a tool covering different domains.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with MoCa (0-30/30, the higher the better cognition) | 2 months
  Cognition will be assessed by the MoCa(0-30/30), a tool covering different domains.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with MoCa (0-30/30, the higher the better cognition) | 4 months
  Cognition will be assessed by the MoCa(0-30/30), a tool covering different domains.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with MoCa (0-30/30, the higher the better cognition) | Baseline
  Cognition will be assessed by the MoCa(0-30/30), a tool covering different domains.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with MoCa (0-30/30, the higher the better cognition) | 2 months
  Cognition will be assessed by the MoCa(0-30/30), a tool covering different domains.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with MoCa (0-30/30, the higher the better cognition) | 4 months
  Cognition will be assessed by the MoCa(0-30/30), a tool covering different domains.
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Katz (6-24/24, the higher, more dependent) | Baseline
  Dependency in basic activities of daily living will be scored on the Katz scale (6-24/24).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Katz (6-24/24, the higher, more dependent) | 2 months
  Dependency in basic activities of daily living will be scored on the Katz scale (6-24/24).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Katz (6-24/24, the higher, more dependent) | 4 months
  Dependency in basic activities of daily living will be scored on the Katz scale (6-24/24).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Katz (6-24/24, the higher, more dependent) | Baseline
  Dependency in basic activities of daily living will be scored on the Katz scale (6-24/24).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Katz (6-24/24, the higher, more dependent) | 2 months
  Dependency in basic activities of daily living will be scored on the Katz scale (6-24/24).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Katz (6-24/24, the higher, more dependent) | 4 months
  Dependency in basic activities of daily living will be scored on the Katz scale (6-24/24).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Lawton (9-27/27, the higher, more independent) | Baseline
  Dependency in instrumental activities of daily living will be scored on Lawton scale (9-27/27).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Lawton (9-27/27, the higher, more independent) | 2 months
  Dependency in instrumental activities of daily living will be scored on Lawton scale (9-27/27).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Lawton (9-27/27, the higher, more independent) | 4 months
  Dependency in instrumental activities of daily living will be scored on Lawton scale (9-27/27).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Lawton (9-27/27, the higher, more independent) | Baseline
  Dependency in instrumental activities of daily living will be scored on Lawton scale (9-27/27).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Lawton (9-27/27, the higher, more independent) | 2 months
  Dependency in instrumental activities of daily living will be scored on Lawton scale (9-27/27).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in functional ability measured with Lawton (9-27/27, the higher, more independent) | 4 months
  Dependency in instrumental activities of daily living will be scored on Lawton scale (9-27/27).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in quality of life (Qol) measured with SarQol (short form, 14 items: 4-point Likert Scale: 0-100/100, the higher, the better Qol) | Baseline
  Qol will be scored on SarQol (short form, 14 items: 0-100/100, the higher, the better Qol)
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in Qol measured with SarQol (short form, 14 items: 4-point Likert Scale: 0-100/100, the higher, the better Qol) | 2 months
  Qol will be scored on SarQol (short form, 14 items: 0-100/100, the higher, the better Qol)
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in Qol measured with SarQol (short form, 14 items: 4-point Likert Scale: 0-100/100, the higher, the better Qol) | 4 months
  Qol will be scored on SarQol (short form, 14 items: 0-100/100, the higher, the better Qol)
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in Qol measured with SarQol (short form, 14 items: 4-point Likert Scale: 0-100/100, the higher, the better Qol) | Baseline
  Qol will be scored on SarQol (short form, 14 items: 0-100/100, the higher, the better Qol)
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in Qol measured with SarQol (short form, 14 items: 4-point Likert Scale: 0-100/100, the higher, the better Qol) | 2 months
  Qol will be scored on SarQol (short form, 14 items: 0-100/100, the higher, the better Qol)
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in Qol measured with SarQol (short form, 14 items: 4-point Likert Scale: 0-100/100, the higher, the better Qol) | 4 months
  Qol will be scored on SarQol (short form, 14 items: 0-100/100, the higher, the better Qol)
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in Qol measured with Eq-5D-5L (0 no problem, 5 extreme problems + visual analogue scale(VAS) 0-100/100, the higher the better Qol). | Baseline
  Qol will be scored on Eq-5D-5L(0-35 & VAS 0 (worst Qol) to 100 (best Qol)).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in Qol measured with Eq-5D-5L (0 no problem, 5 extreme problems + visual analogue scale(VAS) 0-100/100, the higher the better Qol). | 2 months
  Qol will be scored on Eq-5D-5L(0-35 & VAS 0 (worst Qol) to 100 (best Qol)).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the changes in intrinsic capacity as measured with ISHA and the changes in Qol measured with Eq-5D-5L (0 no problem, 5 extreme problems + visual analogue scale(VAS) 0-100/100, the higher the better Qol). | 4 months
  Qol will be scored on Eq-5D-5L(0-35 & VAS 0 (worst Qol) to 100 (best Qol)).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in Qol measured with Eq-5D-5L (0 no problem, 5 extreme problems + visual analogue scale(VAS) 0-100/100, the higher the better Qol). | Baseline
  Qol will be scored on Eq-5D-5L(0-35 & VAS 0 (worst Qol) to 100 (best Qol)).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in Qol measured with Eq-5D-5L (0 no problem, 5 extreme problems + visual analogue scale(VAS) 0-100/100, the higher the better Qol). | 2 months
  Qol will be scored on Eq-5D-5L(0-35 & VAS 0 (worst Qol) to 100 (best Qol)).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)
The correlation between the variability in intrinsic capacity as measured with ISHA and the changes in Qol measured with Eq-5D-5L (0 no problem, 5 extreme problems + visual analogue scale(VAS) 0-100/100, the higher the better Qol). | 4 months
  Qol will be scored on Eq-5D-5L(0-35 & VAS 0 (worst Qol) to 100 (best Qol)).
  Vitality capacity:
  Maximal grip strength(kPa) Respiratory muscle strength(cmH2O) Muscle fatigue resistance(s) Self-perceived fatigue questionnaire(Question(Q) 1: 1 Not tired, 7 Extremely tired; Q2: 1 No I don't agree, 7 Yes I agree & MFI: 0 Not fatigue, 5 Fatigue)
  Locomotor capacity:
  Timed up and go(s) 4-meter gait speed(m/s) Balance test(progressive standing: first 2 tests: 0 Impossible, 1 Holding for 10s; last test: 0 Impossible, 1 Holding for >3s-<9s, 2 holding for 10s) 30-second chair stand(n)
  Sensory capacity:
  Hearing test(signal to noise technology) Vision test(rotating E test)
  Cognitive capacity:
  Orientation test(0 Incorrect, 1 Correct) Object naming from description(0 Incorrect, 1 Correct) Verbal fluency(n) 10-words immediate & delayed recall(0 Incorrect, 1 Correct)
  Psychological capacity:
  Resilience questionnaire(1 Strongly disagree, 5 Strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Bautmans, Prof. Dr., Principal Investigator — VUB

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Frailty & resilience in ageing research group VUB site — http://fria.research.vub.be/
- See also: ISHA-AAL site — http://www.aal-europe.eu/projects/isha/